CLINICAL TRIAL: NCT00932711
Title: Limited Intervention in Low Risk(Tier 3) COPD Patients
Brief Title: Effect of Educational Intervention in Patients With Low-Risk Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: VA Midwest Health Care Network (U.S. Federal Agency)
Responsible Party: Kathryn Rice, MD, Minneapolis VA Medical Center
Organization: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4140-B
Record Dates: First submitted 2009-07-02; First posted 2009-07-03 (Estimated); Last update posted 2009-07-03 (Estimated); Status verified 2009-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Educational intervention (Experimental): Subjects in this group will receive educational brochures about management of COPD
  Interventions: Behavioral: Educational brochures

INTERVENTIONS:
Behavioral: Educational brochures — A locally developed educational brochure containing information about smoking cessation, influenza and pneumococcal vaccination, regular exercise, compliance with prescribed COPD therapy and recognition of symptoms, along with a goal setting questionnaire

SUMMARY:
The purpose of this study is to determine if educational intervention is effective in reducing exacerbations of chronic obstructive pulmonary disease in patients with low-risk disease.

DETAILED DESCRIPTION:
There is growing evidence about the effectiveness of case management in preventing adverse events in patients with high-risk chronic obstructive pulmonary disease(COPD). But the majority of COPD patients belong to the low-risk category. We propose that a less intense educational intervention will have a similar beneficial effect in reducing hospital admissions and emergency department (ED) visits in this larger group of low-risk COPD patients.

ELIGIBILITY:
Inclusion Criteria: Spirometrically confirmed COPD in VISN23 registry. FEV1/FVC <70%.

Exclusion Criteria:Hospital admissions or ED visits in the VISN23 disease registry for COPD within last one year

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-06 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Combined frequency of admissions and ED visits for COPD over 1 year. | One year

SECONDARY OUTCOMES:
Patient knowledge of COPD will be compared. | 1 year
Use of respiratory medications will be compared | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Rice, MD, Principal Investigator — Minneapolis Veterans Affairs Medical Center
Locations (1):
- Minneapolis VA Medical Center, Minneapolis, Minnesota, United States